CLINICAL TRIAL: NCT05083559
Title: A Crossover Study to Assess the Efficacy of a Robust AP Closed Loop System vs MPC Closed Loop System
Brief Title: Two Way Crossover Closed Loop Study R-AP vs MPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jessica Castle, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23343; 5R01DK120367-04 (NIH)
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Type 1 Diabetes
Keywords: glucose sensor; automated insulin delivery systems
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MPC AP system (Experimental): Participants will use the MPC AP system for automated insulin delivery for a 9 hour study visit.
  Interventions: Device: MPC AP algorithm
- Robust R-AP system (Experimental): Participants will use the Robust R-AP system for automated insulin delivery for a 9 hour study visit.
  Interventions: Device: Robust R-AP algorithm

INTERVENTIONS:
Device: MPC AP algorithm — The Model Predictive Control (MPC) insulin infusion algorithm contains a model within the controller that takes as an input the aerobic metabolic expenditure in addition to the CGM and meal inputs. The algorithm uses heart rate and accelerometer data collected on the patient's body to calculate metabolic expenditure. The metabolic expenditure then acts on the model for the insulin dynamics, whereby more energy expenditure and longer duration exercise can lead to a more substantial effect of insulin on the CGM.
  Arms: MPC AP system
Device: Robust R-AP algorithm — The R-AP is a modified MPC algorithm. A new feature in the algorithm includes a model for missed meal insulin detection. The model includes estimations for carbohydrate consumption based glucose patterns to determine if that person has consumed a meal without announcing it to the system.
  Arms: Robust R-AP system

SUMMARY:
An artificial pancreas (AP) is a control system for automatic insulin delivery. The investigators have implemented a missed meal bolus detection algorithm for use within an AP control system. The robust R-AP system used in this protocol has been designed to handle a variety of real-world scenarios that are critical to a high-risk patient population. The investigators will test how well the new algorithm handles missed or inaccurate meal announcements. This type of algorithm may significantly improve glucose control over the standard model predictive control (MPC) closed-loop algorithm without these new algorithm features for patients with type 1 diabetes.

DETAILED DESCRIPTION:
Participants will undergo two visits at Oregon Health and Science University (OHSU) that will evaluate missed meal bolus detection. Participants will arrive at approximately 7am for all visits, be monitored through the afternoon and discharged before dinner. During each of these intervention visits, participants will wear an Omnipod to deliver insulin and a Dexcom G6 Continuous Glucose Monitoring System (CGM) to measure glucose. The closed loop system will receive activity data through a Polar M600 watch worn by the participant. The studies will test the ability of the system to adapt to a missed meal bolus. Participants will eat self selected meals at 10 am and 2pm, both meals with a missed bolus, and these meals will be repeated across both study arms. For one missed meal bolus study, glucose will be controlled using the Robust R-AP closed-loop mode. During the other missed meal bolus study, glucose will be controlled using the MPC closed-loop mode. Participants will complete frequent glucose and ketone checks for safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female participants 18 to 65 years of age.
* Current use of an insulin pump for at least 3 months with stable insulin pump settings for >2 weeks.
* HbA1c ≤ 10.5% at screening.
* Total daily insulin requirement is less than 139 units/day.
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intra-uterine device (IUD), the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Renal insufficiency (GFR < 60 ml/min, using the Modification of Diet in Renal Disease (MDRD) equation as reported by the OHSU laboratory).
* Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
* Hematocrit of less than 36% for men, less than 32% for women.
* History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator. Participants will complete a hypoglycemia awareness questionnaire. Participants will be excluded for four or more R responses.
* History of diabetes ketoacidosis during the prior 6 months prior to screening visit, as diagnosed on hospital admission or as judged by the investigator.
* Adrenal insufficiency.
* Any active infection.
* Known or suspected abuse of alcohol, narcotics, or illicit drugs.
* Seizure disorder.
* Active foot ulceration.
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
* Major surgical operation within 30 days prior to screening.
* Use of an investigational drug within 30 days prior to screening.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* Allergy to aspart insulin.
* Current administration of oral or parenteral corticosteroids.
* Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* Beta blockers or non-dihydropyridine calcium channel blockers.
* Current use of any medication intended to lower glucose other than insulin (ex. use of liraglutide).
* Gastroparesis
* Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the participant's safety or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jacobs, PhD, Principal Investigator — Oregon Health and Science University; Jessica Castle, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MPC to R-AP: The randomization order for participants in this arm was Model Predictive Control (MPC) followed by Robust-Artificial Pancreas (R-AP). Each visit was about 8 hours long.
- R-AP to MPC: The randomization order for participants in this arm was Robust-Artificial Pancreas (R-AP followed by Model Predictive Control (MPC). Each visit was about 8 hours long.
Period: Dexcom Training Visit (30 Minutes)
Arm/Group | MPC to R-AP | R-AP to MPC
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: First Rest Period (1-12 Weeks)
Arm/Group | MPC to R-AP | R-AP to MPC
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: First Intervention (~8 Hours)
Arm/Group | MPC to R-AP | R-AP to MPC
Started | 7 | 8
Completed | 3 | 7
Not Completed | 4 | 1
Not completed — hit stopping rules for hyperglycemia | 4 | 1
Period: Second at Home Period (3-30 Days)
Arm/Group | MPC to R-AP | R-AP to MPC
Started | 7 | 8
Completed | 5 | 8
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention Visit (~8 Hours)
Arm/Group | MPC to R-AP | R-AP to MPC
Started | 5 | 8
Completed | 4 | 8
Not Completed | 1 | 0
Not completed — hit stopping rules for hyperglycemia | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MPC to R-AP: The randomization order for participants in this arm was Model Predictive Control (MPC) followed by Robust-Artificial Pancreas (R-AP). Each visit was about 72 hours and included a 12 hour inpatient and 60 hour outpatient portion.
- R-AP to MPC: The randomization order for participants in this arm was Robust-Artificial Pancreas (R-AP followed by Model Predictive Control (MPC). Each visit was about 72 hours and included a 12 hour inpatient and 60 hour outpatient portion.
- Total: Total of all reporting groups
Arm/Group | MPC to R-AP | R-AP to MPC | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (10.1) | 34.1 (9.9) | 37.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Postprandial Glucose
Description: Incremental AUC of postprandial glucose in the 4 hours following the start of first meal. AUC (mg/dL*hr) will be calculated using a trapezoidal method, which sums all CGM values taken every 5 minutes in the 4 hour period following the meal above the starting glucose. This yields a maximum of 48 data points for the calculation.
Time Frame: 4 hour period following the first meal
Measure: Mean (Standard Deviation); unit: mg/dL*hr
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
mg/dL*hr | 277.5 (159.4) | 253.9 (105.9)

2. Primary Outcome: Percent of Time With Sensed Glucose Between 70-180 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values between 70-180 mg/dl using Dexcom sensor for the four hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
percentage of time | 24.3 (20.1) | 33.4 (22.8)

3. Secondary Outcome: Percent of Time With Sensed Glucose <70 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 70 mg/dl using Dexcom sensor for the 4 hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
percentage of time | 0 (0) | 1.7 (6.0)

4. Secondary Outcome: Number of Carbohydrate Treatments
Description: Assess the cumulative number of carbohydrate treatments (defined as 15 or 20 grams of carbohydrate) for the four hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Number; unit: carbohydrate treatments
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
carbohydrate treatments | 0 | 2

5. Secondary Outcome: Number of Provider-administered Insulin Injections
Description: Assess the cumulative number of provider-administered insulin injections to treat hyperglycemia in the 4 hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Number; unit: insulin injections
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
insulin injections | 4 | 2

6. Secondary Outcome: Mean Sensed Glucose
Description: Assess the mean sensed glucose from the Dexcom G6 reported sensor glucose values for the four hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
mg/dL | 230.8 (43.6) | 212.6 (49.6)

7. Secondary Outcome: Percent of Time With Sensed Glucose <54 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 54 mg/dl using Dexcom sensor for the four hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
percentage of time | 0 (0) | 0.8 (2.7)

8. Secondary Outcome: Percent of Time With Sensed Glucose >180 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values greater than 180 mg/dl using Dexcom sensor for the four hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
percentage of time | 75.7 (20.2) | 64.8 (24.1)

9. Secondary Outcome: Percent of Time With Sensed Glucose >250 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values greater than 250 mg/dl using Dexcom sensor for the four hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
percentage of time | 36.9 (26.5) | 31.6 (26.0)

10. Secondary Outcome: Mean Amount of Insulin Delivered Per Day (in Units)
Description: Assess the mean amount of insulin delivered per day by the Omnipod through the AP system study in units for the four hour period following the first meal.
Time Frame: 4 hour period following the first meal
Measure: Mean (Standard Deviation); unit: units
Arm/Group | MPC AP System | Robust R-AP System
Number analyzed (Participants) | 13 | 13
units | 7.6 (3.3) | 8.7 (3.2)

ADVERSE EVENTS:
Time Frame: 3 months
Description: All participants that began/started the Dexcom training visit or a MPC or R-AP arm are included in the adverse events. The numbers from the participant flow indicate that 15 subjects began the Dexcom training visit, 15 subjects began an MPC visit and 15 subjects began an R-AP visit.
Arm/Group | MPC AP System | Robust R-AP System
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 1/15 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPC AP System (N=15) | Robust R-AP System (N=13)
High ketones (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Blood ketones were measured at 3.4 mmol/L using Precision Xtra ketone meter. Patient was asymptomatic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT05083559/Prot_SAP_000.pdf